CLINICAL TRIAL: NCT00369655
Title: Phase II Trial of VEGF Trap in Patients With Metastatic Breast Cancer Previously Treated With Anthracycline and/or Taxane
Brief Title: VEGF Trap in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01827; NCCTG-N0537; U10CA025224 (NIH); CDR0000491314 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Results first posted 2014-05-05 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2013-11

CONDITIONS: Metastatic Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — aflibercept

ARMS (1):
- Treatment (ziv-afibercept) (Experimental): Patients receive VEGF Trap IV over 1 hour on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: ziv-aflibercept

INTERVENTIONS:
Biological: ziv-aflibercept
  Other Names: aflibercept; vascular endothelial growth factor trap; VEGF Trap; Zaltrap

SUMMARY:
This phase II trial is studying how well VEGF Trap works in treating patients with metastatic breast cancer. VEGF Trap may stop the growth of tumor cells by blocking blood flow to the tumor

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the antitumor activity of VEGF Trap, in terms of tumor response rate, in patients with metastatic breast cancer who have received =< 2 prior chemotherapy regimens for metastatic disease, including a taxane and/or anthracycline.

II. Assess the 6-month progression-free survival rate in patients treated with VEGF Trap.

SECONDARY OBJECTIVES:

I. Describe the adverse event profile (grade using the NCI CTCAE version 3.0) of VEGF Trap in these patients.

II. Describe the progression-free survival times in patients treated with VEGF Trap.

III. Describe the overall survival of patients treated with VEGF Trap. IV. Describe the duration of response in patients treated with VEGF Trap.

OUTLINE: This is a multicenter study.

Patients receive VEGF Trap IV over 1 hour on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3-6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the breast

  * Clinical evidence of metastatic disease
* No more than 2 prior chemotherapy regimens for metastatic disease

  * Prior neoadjuvant or adjuvant chemotherapy allowed*
  * At least 1 prior regimen (in any setting) must have included a taxane and/or an anthracycline
* Measurable disease, defined as ≥ 1 lesion whose longest diameter can be accurately measured per RECIST criteria

  * No nonmeasurable disease, defined as all other lesions, including small lesions(longest diameter < 20 mm) and truly nonmeasurable lesions, including the following:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Inflammatory breast disease
    * Lymphangitis cutis/pulmonis
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesions
* Patients with HER2-positive tumors (3+ by immunohistochemistry or amplified by fluorescent in situ hybridization [FISH]) must have received ≥ 1 prior trastuzumab (Herceptin®)-containing regimen in either the adjuvant or metastatic setting, unless there was a contraindication
* No known CNS metastases
* No evidence of leptomeningeal involvement
* Hormone receptor status not specified
* Male or female
* Menopausal status not specified
* ECOG performance status 0-1
* Life expectancy > 3 months
* WBC ≥ 3,000/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 75,000/mm³
* Hemoglobin > 8.0 g/dL
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 3 times ULN
* AST and ALT ≤ 2.5 times ULN
* Creatinine ≤ 1.5 times ULN
* Urine protein:creatinine ratio < 1 OR urine protein < 500 mg by 24-hour urine collection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after completion of study treatment
* No significant traumatic injury within the past 4 weeks
* No history of allergy or hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies, drug product excipients, or agents chemically or biologically similar to VEGF Trap
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 28 days
* No nonhealing wound, fracture, or ulcer
* No stage III or IV invasive, nonbreast malignancy within the past 5 years
* No history of lung carcinoma of squamous cell type
* No clinically significant cardiovascular disease, including any of the following:

  * Cerebrovascular accident or stroke within the past 6 months
  * Uncontrolled hypertension, defined as blood pressure (BP) > 150/100 mm Hg OR systolic BP > 180 mm Hg if diastolic blood pressure < 90 mm Hg on ≥ 2 separate occasions within the past 3 months
  * Myocardial infarction, coronary artery bypass graft, or unstable angina within the past 6 months
  * New York Heart Association class III or IV cardiovascular disease
  * Serious cardiac arrhythmia requiring medication
  * Peripheral vascular disease ≥ grade 2 within the past 6 months
  * Pulmonary embolism, deep vein thrombosis, or other thromboembolic event within the past 6 months
* No evidence of bleeding diathesis or uncontrolled coagulopathy
* No active, unresolved infection
* No serious concurrent medical condition that would preclude study participation
* No other condition or circumstance that would preclude compliance with study requirements
* See Disease Characteristics
* Prior hormonal therapy in the neoadjuvant, adjuvant, or metastatic setting allowed
* No prior bevacizumab
* More than 4 weeks since prior chemotherapy, endocrine therapy, experimental drug therapy, or immunotherapy and recovered
* More than 4 weeks since prior major surgery or open biopsy
* More than 7 days since prior core biopsy
* More than 2 weeks since prior radiotherapy, except if to a nontarget lesion only

  * Prior radiotherapy to a target lesion allowed only if there has been clear progression of the lesion since radiotherapy was completed
  * Prior single-dose palliative radiotherapy within the past 2 weeks allowed
* No concurrent major surgery
* No concurrent trastuzumab
* Concurrent full-dose anticoagulants (e.g., warfarin) with PT INR > 1.5 allowed provided the following criteria are met:

  * INR in-range (usually between 2 and 3) on a stable dose of oral anticoagulant or on a stable dose of low molecular weight heparin
  * No active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices)
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent participation in another investigational clinical trial
* No other concurrent chemotherapeutic agents, endocrine therapy, biologic agents, radiotherapy, or other nonprotocol antitumor therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-01; Primary Completion 2008-03 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edith Perez, Principal Investigator — North Central Cancer Treatment Group
Locations (1):
- North Central Cancer Treatment Group, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-one women were enrolled during the first stage of the study between January 2007 and March 2008.
Period: Overall Study
Arm/Group | Treatment (Ziv-afibercept)
Started | 21
Completed | 19
Not Completed | 2
Not completed — Refusal of further treatment | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ziv-afibercept)
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 58 [34 to 75]
Sex/Gender, Customized [Number; unit: participants]
  Female | 21
Region of Enrollment [Number; unit: participants]
  United States | 21
ECOG Performance Score [Number; unit: Participants] — The Eastern Cooperative Oncology Group (ECOG) score classified patients according to their functional impairment. Scores range from 0 (fully active) to 5 (death).
  Participants
    0-Fully active | 14
    1-Ambulatory, restricted strenuous activity | 7
Cell type [Number; unit: Participants]
  Infiltrating ductal | 16
  Infiltrating lobular | 1
  Comedo | 1
  Inflammatory | 1
  Infiltrating ductal and comedo | 1
  Missing | 1
Dominant Disease [Number; unit: Participants]
  Visceral | 15
  Nonvisceral | 6
Visceral Disease Site [Number; unit: Participants] — The presented results are for the 15 participants with visceral disease. The same participant may report more than one disease site.
  Participants
    Liver | 7
    Lung | 7
    Abodomen | 1
    Other | 2
Estrogen Receptor (ER) Result [Number; unit: Participants]
  Positive | 9
  Negative | 12
Progesterone Receptor (PR) Result [Number; unit: Participants]
  Positive | 5
  Negative | 16
Human epidermal growth factor receptor 2 (HER2) Result [Number; unit: Participants]
  Positive | 4
  Negative | 14
  HER2 testing not done | 3
Previous (Neo) Adjuvant Chemotherapy [Number; unit: Participants]
  Yes | 13
  No | 8
Number of Previous Chemotherapy Regimens [Number; unit: Participants]
  0 | 3
  1 | 11
  2 | 7
Previous Hormonal Therapy [Number; unit: Participants]
  Yes | 9
  No | 12
Previous Trastuzumab [Number; unit: Participants]
  Yes | 5
  No | 16
Prior Anthracyclines [Number; unit: Participants]
  Yes | 15
  No | 6
Prior Taxanes [Number; unit: Participants]
  Yes | 19
  No | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Confirmed Tumor Response
Description: Confirmed tumor response was defined as the total number of efficacy-evaluable patients who achieved a complete or partial response according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria on 2 consecutive evaluations at least 8 weeks apart.
Time Frame: Up to 5 years
Population: All participants who have met the eligibility criteria, who have signed a consent form and have begun treatment were evaluable for response.
Measure: Number; unit: Participants
Arm/Group | Treatment (Ziv-afibercept)
Number analyzed (Participants) | 21
Participants
  Confirmed tumor partial response | 1
  No Confirmed reponse | 20

2. Primary Outcome: Proportion of Patients Receiving Vascular Endothelial Growth Factor (VEGF) Trap With 6-month Progression-free Survival
Description: The 6-month progression free survival rate was defined as the proportion of efficacy-evaluable patients on study treatment and progression-free 6 months from registration. Patients who died without documentation of progression will be considered to have progressed on the date of their death.
Time Frame: 6 months
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Treatment (Ziv-afibercept)
Number analyzed (Participants) | 21
Participants | 2

3. Secondary Outcome: Progression Free Survival
Description: Progression-free survival was defined as the number of months from registration to the date of disease progression or death, with patients who died without documentation of progression being considered to have progressed on the date of their death.
Time Frame: Time from registration to disease progression or death (up to 5 years)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Ziv-afibercept)
Number analyzed (Participants) | 21
Months | 2.7 [1.8 to 5.0]

4. Secondary Outcome: Overall Survival
Description: Overall survival time was defined as the number of months from registration to the date of death or last follow-up
Time Frame: Time from registration to death or last follow up (up to 5 years)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Ziv-afibercept)
Number analyzed (Participants) | 21
Months | 12.7 [6.7 to 31.1]

5. Secondary Outcome: Median Duration of Response
Description: Duration of response was defined as for all evaluable patients who have achieved an objective response as the date at which the patient's objective status is first noted to be either a complete response or partial response to the date progression is documented.
Time Frame: Up to 5 years
Population: Analysis population included only patients who have achieved a confirmed tumor response. The duration of response of 4.6 months is reported from one patient.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Ziv-afibercept)
Number analyzed (Participants) | 1
Months | 4.6 [4.6 to 4.6]

6. Secondary Outcome: Number of Participant With Previous Treatment of Anti-HER2 With Cardiac Events
Time Frame: Up to 5 years
Population: All participants who have received previous treatment with anti-HER2.
Measure: Number; unit: Participants
Arm/Group | Treatment (Ziv-afibercept)
Number analyzed (Participants) | 5
Participants | 1

ADVERSE EVENTS:
Time Frame: Start of treatment to end of treatment
Description: Common Toxicity Criteria for Adverse Events (CTCAE) v3
Arm/Group | Treatment (Ziv-afibercept)
Serious Adverse Events (participants affected / at risk) | 10/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ziv-afibercept) (N=21)
Left ventricular failure (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ziv-afibercept) (N=21)
Hemoglobin decreased (Blood and lymphatic system disorders) | 2 (2)
Flashing vision (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 3 (6)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 11 (25)
Diarrhea (Gastrointestinal disorders) | 12 (19)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 2 (3)
Mucositis oral (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 11 (23)
Vomiting (Gastrointestinal disorders) | 9 (14)
Chest pain (General disorders) | 9 (22)
Fatigue (General disorders) | 21 (75)
Pain (General disorders) | 2 (2)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (6)
Alkaline phosphatase increased (Investigations) | 6 (10)
Aspartate aminotransferase increased (Investigations) | 4 (13)
Bilirubin increased (Investigations) | 2 (3)
INR increased (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 4 (7)
Neutrophil count decreased (Investigations) | 2 (3)
Platelet count decreased (Investigations) | 1 (1)
Weight loss (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 9 (17)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 8 (13)
Joint pain (Musculoskeletal and connective tissue disorders) | 13 (26)
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (21)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 9 (23)
Memory impairment (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (3)
Proteinuria (Renal and urinary disorders) | 5 (9)
Urethral pain (Renal and urinary disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (15)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 13 (44)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (4)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 3 (4)
Hypertension (Vascular disorders) | 12 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less